CLINICAL TRIAL: NCT01763489
Title: Impact of a Graphical Tool on the Reader's Interpretation of Surgical RCT Applicability In the Field of Digestive Cancer
Brief Title: ASSIST Tool and Surgical Randomized Controlled Trial Applicability
Acronym: ASTA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Isabelle BOUTRON, Professor, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RAV004
Record Dates: First submitted 2013-01-03; First posted 2013-01-09 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Digestive Cancer
Keywords: randomized controlled trial; applicability; ASSIST tool; surgery; digestive cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASSIST tool group (Experimental): Surgeons will assess the applicability of a trial using the ASSIST
  Interventions: Behavioral: Applicability Assessment
- Synopsis Group (Active Comparator): Surgeons will assess the applicability of a trial using the synopsis presented in a case vignette
  Interventions: Behavioral: Applicability Assessment

INTERVENTIONS:
Behavioral: Applicability Assessment — assess the applicability of a trial using the ASSIST tool or the synopsis

SUMMARY:
Background: The ASSIST tool is a graphical tool to represent and evaluate the applicability of a surgery trial to improve the translation of research to practice.

Objective: To evaluate the impact of the ASSIST tool on the interpretation of the applicability of randomized controlled trials (RCTs) in the field of digestive cancer surgery.

Design: This study is a randomized controlled trial with two parallel arms. Participants: Surgeons who contribute to the assessment of manuscripts as experts (peer-reviewer) for international scientific journals of surgery (Annals of Surgery, Archives of Surgery, Gastrointestinal Surgery World Journal of International Journal of Surgical Oncology).

Intervention: Surgeons will be randomized into 2 groups. A group that will evaluate a case vignette (synopsis) of a randomized trial in surgery, and the other group that will evaluate the same case vignette with the representation of the external validity of the trial with ASSIST tool.

Outcome measures: Participants will indicate on a numeric scale range from 1 to 10 if they feel able to judge the applicability of the trial for 1) patients, 2) centers, 3) surgeons and 4) intervention.

Sample Size: 28 case vignettes with randomized trials and their ASSIST tool have been developed and evaluated. The inclusion of 130 participants (65 per arm) is required.

DETAILED DESCRIPTION:
The study will be conducted in 2 steps:

In a first step, investigators will develop cases vignettes of published RCTs evaluating surgical interventions in the field of digestive cancer with its representations of external validity according to ASSIST.

In a second step, investigators will invite a panel of peer reviewers to appraise the external validity (applicability) of selected RCTs without and with the graphical tool (ASSIST), on a security web site.

ELIGIBILITY:
Inclusion Criteria:

* surgeons
* who contribute to the assessment of manuscripts as experts (peer-reviewer) for international scientific journals of surgery (Annals of Surgery, Archives of Surgery, Gastrointestinal Surgery World Journal of International Journal of Surgical Oncology)

Exclusion Criteria:

* No one

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
feeling able to judge the applicability of the trial | 2 months
  Participants will indicate on a numeric scale range from 1 to 10 if they feel able to judge the applicability of the trial for patients

CONTACTS AND LOCATIONS:
Overall Officials: Boutron Isabelle, Principal Investigator — Assistance Publique - Hôpitaux de Paris